CLINICAL TRIAL: NCT06349356
Title: " Prospective Evaluation of Efficacy and Safety of C.STIM® , an Intense Pulsed Light Device to Treat Signs and Symptoms of Dry Eye Disease (DED)"
Brief Title: Prospective Evaluation of Efficacy and Safety of an Intense Pulsed Light Device to Treat Dry Eye Disease"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quantel Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FDACSTIM0012023; IRB00000533 (Other: WCG IRB)
Record Dates: First submitted 2024-03-22; First posted 2024-04-05 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-05

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: MULTI-CENTER, PROSPECTIVE, RANDOMIZED, SHAM-CONTROLLED, SUPERIORITY, NON-SIGNIFICANT RISK
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intense Pulsed Light treated arm (Experimental): The treatment consists in Intense Pulsed Light C.STIM® with recommended fluence.
  Interventions: Device: Intense pulsed light with C.STIM device
- Very low fluence Intense Pulsed Light arm (placebo) (Placebo Comparator): The treatment consists in Intense Pulsed Light C.STIM® with a very low fluence.
  Interventions: Device: Intense pulsed light with C.STIM device

INTERVENTIONS:
Device: Intense pulsed light with C.STIM device — 4 flashes per treatment session

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of C.STIM, an intense pulsed light device to treat signs and symptoms of dry eye disease. The main question it aims to answer is:

• Difference of the evolution of Tear Break-Up time (TBUT) between the 2 arms of the study (placebo and treated).

Researchers will compare treated group and placebo to respond to the main question.

Participants will assess to an inclusion visit (disease evaluation purpose) and then four IPL treatment visit to finish with the last visit (disease evaluation purpose).

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to read, understand and sign an information consent and image right forms
* aged over 22 years old
* Fitzpatrick skin type I-IV
* Patient is able and willing to comply with the treatment/FU schedule and requirements
* Meibomian Gland Score : Meibum Quality according to Tear Film and Occular Surface Society recommendation: ≥ 16 for 1 eye and 8 central glands in the lower eyelid
* At least 5 non-atrophied meibomian glands in the lower eyelid
* Tear break-up time (TBUT) ≤ 10 seconds
* Symptoms self-assessed using the Occular Surface Disease Index questionnaire ≥ 23

Exclusion Criteria:

* Fitzpatrick skin type V or VI
* Contact lens wear within the month prior to screening
* Unwilling to discontinue use of contact lenses for the duration of the study
* Ocular surgery or eyelid surgery within 6 months prior to screening
* Neuro-paralysis in the planned treatment area within 6 months prior to screening
* Other uncontrolled eye disorders affecting the ocular surface, for example active allergies
* Current use of punctal plugs
* Pre-cancerous lesions, skin cancer or pigmented lesions in the planned treatment area Uncontrolled infections or uncontrolled immunosuppressive diseases
* Patients with ocular infections, within 6 months prior to screening
* Prior history of cold sores or rashes in the perioral area or in the planned treatment area that could be stimulated by light at a wavelength of 610 nm to 1200 nm, including: Herpes simplex 1 & 2, Systemic Lupus erythematosus, and porphyria
* Within 3 months prior to screening, use of photosensitive medication and/or herbs that may cause sensitivity to 610-1200 nm light exposure, including: Isotretinoin, Tetracycline, Doxycycline, and St. John's Wort
* Over exposure to sun, within 4 weeks prior to screening
* Using of topical drops, only artificial tears and glaucoma treatments are authorized
* Radiation therapy to the head or neck, within 12 months prior to screening
* Planned radiation therapy, within 8 weeks after the last treatment session
* Treatment with chemotherapeutic agent, within 8 weeks prior to screening
* Planned chemotherapy, within 8 weeks after the last treatment session
* New topical treatments within the area to be treated (face), or oral therapies, within 3 months prior to screening, analgesics for pain management, oral omega 3 fatty acid supplements are authorized
* Change in dosage of any systemic medication, within 3 months prior to screening
* Anticipated relocation or extensive travel outside of the local study area preventing compliance with follow-up over the study period
* Legally blind in either eye
* History of migraines, seizures or epilepsy
* Facial Itense Pulsed Light treatment, within 12 months prior to screening
* Any thermal treatment of the eyelids, including Lipiflow, within 6 months prior to screening
* Expression of the meibomian glands, within 6 months prior to screening
* In either eye, moderate to severe (Grade 3-4 on the EFRON scale) inflammation of the conjunctiva, including: allergic, vernal or giant papillary conjunctivitis
* In either eye, severe (Grade 4 on the EFRON scale) inflammation of the eyelid, including: blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis
* Ocular surface abnormality that may compromise corneal integrity in either eye (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, or map dot fingerprint dystrophy and pterigyum)
* Eyelid abnormalities that affect lid function in either eye, including: entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, and severe ptosis
* Any systemic condition that may cause dry eye disease, including: Stevens-Johnson syndrome, vitamin A deficiency, rheumatoid arthritis, Wegener's granulomatosis, sarcoidosis, leukemia, Riley-Day syndrome, systemic lupus erythematosus, and Sjögren's syndrome
* Unwilling or unable to abstain from the use of medications known to cause dryness (e.g., isotretinoin, antihistamines) throughout the study duration. Patients must discontinue these medications for at least 1 month prior to the baseline visit.
* Any condition revealed whereby the investigator deems the Patient inappropriate for this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Tear Break-Up Time evolution | 60 days
  Difference of the evolution of Tear Break-Up time (TBUT) between the 2 arms of the study (placebo and treated).

SECONDARY OUTCOMES:
dry eye signs and symptoms | 60 days
  Evolution of dry eye signs and symptoms: DEQ5, Dry Eye Questionnaire 5, score varies from 0 (normal) to 22 (severe symptoms).
dry eye signs and symptoms | 60 days
  Evolution of dry eye signs and symptoms: NIBUT, Non Invasive Break Up Time, normal if higher than 10 second.
dry eye signs and symptoms | 60 days
  Evolution of dry eye signs and symptoms: OSDI, the Ocular Surface Disease Index is a questionnaire with score from 0 (normal) to 100 (severe dry eye symptoms)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 60 days
  Assessment of device safety and tolerability (ocular and dermatologic aspect) : comparison of number of adverse event occurence between the two arms
Meibum quality | 60 days
  Quality of meibum evaluation by Meibomian gland secretion assessment using Meibum Quality : : is assessed in each of 8 glands of the central third of the lower lid on a 0-3 scale for each gland: 0=clear meibum / 1=cloudy meibum/ 2=cloudy with debris (granular)/3=thick, like toothpaste
Meibum Expressibility | 60 days
  Quality of meibum evaluation by Meibomian gland secretion assessment using Meibum Expressibility : Expressibility of meibum is assessed from 5 glands:
  0= all glands expressible / 1=3-4 glands expressible/ 2= 1-2 glands expressible./ 3=no glands expressible.
Use of artificial tear drops | 60 days
  Change in use of artificial tear drops frequency before treatment and after treatment
Use of artificial tear drops | 60 days
  Change in use of artificial tear drops quantity before treatment and after treatment
Glaucoma | 60 days
  Observation of the difference in evolution of dry eye disease in glaucoma vs non-glaucoma patients : comparaison of the Tear Break Up Time in second (normal if superior to 10 seconds)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Visionary Consultants Inc., Lexington, Kentucky
  - Triangle Eye Consultants, Raleigh, North Carolina
  - Toyos Clinic, Nashville, Tennessee
  - Eye Centers of Racine & Kenosha, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No